CLINICAL TRIAL: NCT02272413
Title: A Multicenter, Randomized, Double-blind Phase III Trial to Evaluate Efficacy and Safety of BI 695502 Plus Chemotherapy Versus Avastin® Plus Chemotherapy in Patients With Advanced Nonsquamous Non-Small Cell Lung Cancer
Brief Title: Phase III Trial BI 695502 Plus Chemotherapy vs. Avastin® Plus Chemotherapy in Patients With Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1302.5; 2014-002161-30 (EudraCT Number)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BI 695502 (Experimental)
  Interventions: Drug: BI 695502
- Avastin (Active Comparator)
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: BI 695502
  Arms: BI 695502
Drug: Avastin
  Arms: Avastin

SUMMARY:
The objective of this phase III trial is to establish statistical equivalence in terms of efficacy (best overall response rate [ORR], proportion of patients with complete response [CR] plus partial response [PR]) until 18 weeks of first-line treatment with BI 695502 plus chemotherapy versus Avastin® plus chemotherapy followed by maintenance monotherapy with either BI 695502 or Avastin®.

ELIGIBILITY:
Inclusion criteria:

Adult patients aged >=18 years with histologically or cytologically confirmed advanced nonsquamous non-small cell lung cancer (nsNSCLC). Mixed tumors should be categorized according to the predominant histology.

Note: NSCLC should be predominantly nonsquamous. Recurrent or metastatic disease (Stage IV) with an indication for therapy with paclitaxel + carboplatin + Avastin®.

Patients harboring tumors with unknown or without activating epidermal growth factor receptor (EGFR) / anaplastic lymphoma receptor tyrosine kinase (ALK) mutation maybe included provided chemotherapy is standard of care. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 based on independent central review.

Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.

Adequate hepatic, renal, and bone marrow function:

Life expectancy > 6 months based on clinical judgment. Further inclusion criteria apply.

Exclusion criteria:

Prior therapy with monoclonal antibodies or small molecule inhibitors against Vascular Endothelial Growth Factor (VEGF) or VEGF receptors, including Avastin®.

Prior systemic therapy for metastatic disease. Prior systemic anticancer therapy or radiotherapy for locally advanced nsNSCLC if completed <12 months prior to Screening.

Previous malignancy other than NSCLC in the last 5 years except for basal cell cancer of the skin or pre-invasive cancer of the cervix.

Symptomatic brain metastasis. Diagnosis of small cell carcinoma of the lung, squamous cell carcinoma of the lung, NSCLC not specified (NS) or NSCLC not otherwise specified(NOS).

Any unresolved toxicity > Common Toxicity Criteria Grade 1 (except alopecia) from previous anticancer therapy (including radiotherapy).

History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding. Thrombotic or hemorrhagic event =< 6 months prior to Screening. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (189):
- United States (9):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Lalita Pandit, M.D., Inc., Fountain Valley, California
  - Southern California Oncology Research Alliance, Los Angeles, California
  - Innovative Clinical Research, Inc., Whittier, California
  - Ashland Bellefonte Cancer Center, Ashland, Kentucky
  - Reliant Medical Group, Worcester, Massachusetts
  - Detroit Clinical Research Center, Owosso, Michigan
  - Carolinas Cancer Care, Charlotte, North Carolina
- Argentina (4):
  - CENIT - Centro de Neurociencias, Investigacion y Tratamiento, Ciudad Autonoma Buenos Aires
  - Sanatorio Delta, Rosario
  - Sanatorio Parque, Rosario
  - Centro Oncológico de Rosario, Rosario
- Brazil (13):
  - CPCO - Centro de Pesquisa Clinica em Oncologia, Cachoeiro de Itapemirim
  - Hospital do Cancer do Ceara, Fortaleza
  - Pronutrir, Fortaleza
  - Hospital de Carida de de Ijui - CACON, Ijuí
  - Hospital Bruno Born, Lajeado
  - Hospital da Cidade de Passo Fundo, Passo Fundo
  - Universidade de Caxias do Sul - IPCEM - Inst. de Pesq.clilni, Petrópolis
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André
  - ICAVC - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo
  - ICESP - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Clinica de Oncologia de Sorocaba, Sorocaba
- Bulgaria (7):
  - MHAT - Dobrich, AD, Dobrich
  - UMHAT Georgi Stranski, Clinic of Paediatrics, Pleven, Pleven
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - DCC 1 - Ruse, EOOD, Rousse
  - MHAT Serdika, EOOD, Sofia, Sofia
  - MHAT 'Tokuda Hospital Sofia', EAD, Sofia
  - SHATOD 'Dr. Marko Antonov Markov'-Varna, EOOD, Varna
- Chile (5):
  - Clínica Santa María, Santiago
  - Hospital Clínico San Borja Arriarán, Santiago
  - Centro Internacional de Estudios Clinicos - CIEC, Santiago
  - Instituto Clínico Oncológico del Sur - ICOS, Temuco
  - Hospital Clinico Viña del Mar, Viña del Mar
- Croatia (3):
  - General Hospital Pula, Pula
  - Clinical Hospital Centar Sestre Milosrdnice, Zagreb
  - University Clinic for Pulmonary Diseases, Zagreb
- Egypt (6):
  - Oncology Centre- Mansoura University, Al Mansurah
  - Alexandria University Hospital, Alexandria
  - Ain Shams University Hospital, Cairo
  - National Cancer Institute, Cairo University, Cairo
  - Nasser Institute, Cairo
  - Menofiya University Hospital, Monofia
- Gesundheitszentrum Wetterau gGmbH, Bad Nauheim, Germany
- Greece (6):
  - Athens Hospital of Chest Diseases "Sotiria", Athens
  - University General Hospital of Heraklion, Crete
  - University of Patras Medical School, Pátrai
  - Euromedica Kyanous Stavros General Hospital, Thessaloniki
  - Health Center of Thermi, Thessaloniki, Thessaloniki
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
- Hungary (6):
  - National Koranyi TBC and Pulm. Internal Med. Clinic, Budapest
  - Semmelweis University, Budapest
  - Pulmonology Institute of Veszprem County, Farkasgyepu, Farkasgyepű
  - Jasz-Nagykun-Szolnok Megyei Hetenyi G. Korhaz-Rendelointezet, Szolnok
  - Markusovszky University Teaching Hospital, Szombathely
  - Tudogyogyintezet Torokbalint, Törökbálint
- Italy (4):
  - ASST di Cremona, Cremona
  - Osp. Umberto I, Lugo (RA)
  - Istituto Scientifico Romagnolo, Meldola (FC)
  - Azienda Ospedaliera Universitaria Pisana, Pisa
- Japan (27):
  - Aichi Medical University Hospital, Aichi, Nagakute
  - Aichi Cancer Center Aichi Hospital, Aichi, Okazaki
  - Tosei General Hospital, Aichi, Seto
  - Fujita Health University Hospital, Aichi, Toyoake
  - Aso Co.,Ltd Iizuka Hospital, Fukuoka, Iizuka
  - Gunma Prefectural Cancer Center, Gunma, Ota
  - Hyogo Prefectural Amagasaki General Medical Center, Hyogo, Amagasaki
  - Itami City Hospital, Hyogo, Itami
  - Kobe City Medical Center General Hospital, Hyogo, Kobe
  - Ibaraki Prefectural Central Hospital, Ibaraki, Kasama
  - Kagawa Rosai Hospital, Kagawa, Marugame
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Yokohama City University Hospital, Kanagawa, Yokohama
  - Uji-Tokushukai Medical Center, Kyoto, Uji
  - Matsusaka City Hospital, Mie, Matsusaka
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki, Miyazaki
  - Nara Hospital Kinki University Faculty of Medicine, Nara, Ikoma
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Osaka, Hirakata
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Osaka
  - Takatsuki Red Cross Hospital, Osaka, Takatsuki
  - Saitama Medical University International Medical Center, Saitama, Hidaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakaishi
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
  - Japan Anti-Tuberculosis Association Fukujuji Hospital, Tokyo, Kiyose
  - Toranomon Hospital, Tokyo, Minato-ku
- Malaysia (3):
  - Hospital Pulau Pinang, Georgetown Pulau Pinang
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
- Mexico (6):
  - Investigacion Biomedica para el Desarrollo de Farmacos, El Salto
  - Unidad de Atencion Medica e Investigacion en Salud S.C., Mérida
  - Axis Heilsa S. de R.L. de C.V., Monterrey, Monterrey
  - Clinical Medical Research S.C, Orizaba
  - Hospital San Jose Querétaro, Querétaro
  - Centro Hemato Oncológico Privado, Toluca
- Philippines (5):
  - Dr. Pablo O. Torre Memorial Hospital, Bacolod City
  - Cebu Doctors Hospital, Cebu City
  - Perpetual Succour Hospital (Cebu), Cebu City
  - Manila Doctors Hospital, Manila
  - Lung Center of the Philippines, Quezon City
- Poland (6):
  - Wojewodzkie Centrum Szpitalne Kotliny Jeleniogorskiej, Jelenia Góra
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Zofia Tarnowska domo Zamoyska,RegHosp.Cardiol.Dep,Tarnobrzeg, Tarnobrzeg
  - The Provincial Polyclinical Hospital in Torun, Torun
  - Onco.Cent. - Instit. of Maria Sklodowskiej-Curie, Warsaw
  - Magodent Sp. Z o.o., Warsaw
- Portugal (5):
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Centro Hospitalar Lisboa Norte Hospital Pulido Valente, Lisbon
  - IPO Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E. - Hospital de São Sebastião, Santa Maria da Feira
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Romania (5):
  - Baia Mare Emergency County Hospital, Baia Mare
  - Institute of Oncology 'Prof. Dr. Alexandru Trestioreanu', Bucharest
  - Spitalul Militar de Urgenta Dr.Papilian, Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - S.C Oncocenter Oncologie Clinica S.R.L, Timișoara
- Russia (10):
  - SBIH of Arkhangelsk reg. "Arkhangelsk Clin. Onc. Dispensary", Arkhangelsk
  - St.Auton.Heal.Inst."Rep.Clin.Onc.Disp.of MoH of Rep. Tatarstan", Kazan'
  - RBIH "Kursk regional clinical oncology dispensary", Kursk
  - FSBI "N.N Blokhin Med.Res.Cent.Onc."MoH of RF, Moscow
  - BHI of Omsk region - Clinical Oncology Dispensary, Omsk
  - SBIH of Stavropol territory "Pyatigorsk Oncol. Dispensary", Pyatigorsk
  - GUZ Leningradskaya Regional Clin. Hospital, St. Petersburg, Saint Petersburg
  - 1stPavlov St.Med.Univ.St.-Petersburg Res.Inst., Saint Petersburg
  - SPb SBIH "City Clinical Oncological Dispensary", Saint Petersburg
  - FSBI "N.N. Petrov National Medical Research Center of Oncology" of MoH of RF, Saint Petersburg
- Serbia (5):
  - Institute for Oncol & Radiol of Serbia, Clinic f. Med. Onco., Belgrade
  - Clinical Center Bezanijska kosa, Belgrade, Belgrade
  - Clinic of Pulmonary Diseases and Tuberculosis 'Knez Selo', Gornji Matejevac
  - Inst. for Pulm. Diseases of Vojvodine, Clinic f. Pulm. Oncol, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- South Africa (5):
  - GVI Cape Gate Oncology Centre, Cape Town
  - Rondebosch Oncology Centre, Cape Town
  - GVI Oncology Outeniqua Unit, George
  - West Rand Oncology Centre, Johannesburg, Johannesburg
  - Langenhoven Drive Oncology Centre, Port Elizabeth
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, St.Vincent's Hospital, Suwon
- Spain (8):
  - Hospital Infanta Cristina, Badajoz
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Miguel Servet, Zaragoza
- Thailand (6):
  - Songklanagarind Hospital, Hat Yai
  - Ubonratchathani Cancer Hospital, Muang, Muang
  - Udonthani Cancer Hospital, Muang, Muang
  - Maharaj Nakorn Chiang Mai Hospital, Muang
  - Lampang Hospital, Muang
  - Naresuan University Hospital, Muang
- Turkey (Türkiye) (8):
  - Akdeniz University Medical Faculty, Antalya
  - Inonu Uni. Med. Fac., Battalgazi, Battalgazi
  - Dicle University Medical Faculty, Diyarbakır
  - Trakya Universitesi Tip Fakultesi, Edirne
  - Gaziantep University, Gaziantep
  - Bezmi Alem Foundation University Medical Faculty Hospital, Istanbul
  - Yeditepe University Medical School Hospital, Istanbul
  - Fatih University Faculty of Medicince, Istanbul, Istanbul
- Ukraine (16):
  - CTPI Chernihiv Regional Oncological Dispensary, Chernihiv, Chernihiv
  - Munic.Instit."City Clin.Hosp.#4" of Dnipro City Council, Dnipropetrovsk
  - CHI Kharkiv Regional Clinical Oncological Center, Kharkiv
  - Kherson Regional Oncologic Dispensary, Kherson, Kherson
  - Treatment-Diagnostic CTR of Private Enterprise, Kirovohrad, Kirovohrad
  - CI Kryvyi Rih Oncological Dispensary of DRC, Kryvyi Rih, Dnipropetrovsk
  - National Institute of Cancer, Kyiv
  - Medical and Preventive Treatment Inst. Volyn Regional, Lutsk, Lutsk
  - CI of LRC Lviv Onco.Reg.Treat.&Diag.Cent., Lviv
  - Poltava Regional Clinical Oncological Dispensary, Poltava, Poltava
  - Sumy Regional Oncology Center, Sumy
  - CI of TRC Ternopil RC Oncological Dispensary Thoracic Dept, Ternopil
  - Uzhgorod National University, Oncology Centre, Uzhhorod
  - Transcarpathian Reg Clin Oncological Dispensary, Uzhgorod, Uzhhorod
  - Vinnytsia Regional Clinical Oncological Dispensary, Vinnytsia
  - CI Zapor Reg Cl Oncological Dispensary of ZRC, Zhaporizhzhia, Zhaporizhzhia
- United Kingdom (2):
  - Cheltenham General Hospital, Cheltenham
  - Wythenshawe Hospital, Manchester
- Vietnam (2):
  - Can Tho Oncology Hospital, Can Tho
  - Bach Mai hospital, Hanoi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III, randomized, double-blind, multicenter, active comparator, parallel 2-arm trial in patients with advanced non-squamous non-small cell lung cancer (nsNSCLC). From 21December2017, Sponsor recommended, patients to be switched from BI 695502 to reference product Avastin® (commercially available) as soon as it was available at clinical site.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensure that they (the patients) met all strictly implemented inclusion/exclusion criteria. Patients were not to be randomized to trial treatment if any one of the specific entry criteria were violated.
Groups:
- BI 695502: Patients received BI 695502 solution for i.v. infusion, 15 mg/kg bw, every 3 weeks for up to 6 cycles. During the induction cycles, patients also received standard combination chemotherapy consisting of paclitaxel 200 mg/m^2 body surface area (BSA), followed by carboplatin target area under the curve (AUC) 6 mg/mL*min, with adequate pre- and concomitant medication. After Cycle 4 to 6, for responding or stabilized patients, maintenance treatment with BI 695502 monotherapy could be started per the original randomization. Patients then received BI 695502 as a single agent until disease progression, death, withdrawal of consent, unacceptable toxicity, or until the Switch Visit (when each patient was switched to receive commercially available Avastin®), whichever occurred earlier.
- Avastin® US: Patients received US-licensed Avastin® solution for i.v. infusion, 15 mg/kg bw, every 3 weeks for up to 6 cycles. During the induction cycles, patients also received standard combination chemotherapy consisting of paclitaxel 200 mg/m^2 BSA, followed by carboplatin target AUC 6 mg/mL*min, with adequate pre- and concomitant medication.
  After Cycle 4 to 6, for responding or stabilized patients, maintenance treatment with US-licensed Avastin® monotherapy could be started per the original randomization. Patients then received US-licensed Avastin® as a single agent until disease progression, death, withdrawal of consent, unacceptable toxicity, or until the Switch Visit (when each patient was switched to receive commercially available Avastin®), whichever occurred earlier.
Period: Randomized Through Treatment Start
Arm/Group | BI 695502 | Avastin® US
Started (Started are randomized) | 338 (Started for this period) | 333 (Started for this period)
Treated | 335 | 328
Completed (Completed are treated) | 335 | 328
Not Completed | 3 | 5
Not completed — Not treated | 3 | 5
Period: Pre-switch Period
Arm/Group | BI 695502 | Avastin® US
Started (Started are treated) | 335 (Started for this period) | 328 (Started for this period)
Completed | 42 | 46
Not Completed | 293 | 282
Not completed — Adverse Event | 38 | 37
Not completed — Death | 26 | 26
Not completed — Withdrawal by Subject | 27 | 15
Not completed — Physician Decision | 6 | 18
Not completed — Progressive disease | 185 | 173
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Other than listed | 10 | 11
Period: Post-switch Period
Arm/Group | BI 695502 | Avastin® US
Started | 42 (Started for this period) | 46 (Started for this period)
Completed | 0 | 0
Not Completed | 42 | 46
Not completed — Adverse Event | 4 | 4
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Progressive disease | 21 | 21
Not completed — Study terminated by sponsor | 8 | 11
Not completed — Other than listed | 4 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS contained all randomized patients who received at least 1 dose of trial drug and who had a baseline tumor assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695502 | Avastin® US | Total
Number analyzed (Participants) | 335 | 328 | 663
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (9.89) | 61.3 (9.22) | 61.2 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 125 | 246
  Male | 214 | 203 | 417
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 34 | 77
  Not Hispanic or Latino | 284 | 285 | 569
  Unknown or Not Reported | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 64 | 71 | 135
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 258 | 248 | 506
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR), Based on Unconfirmed Response Assessment, as Assessed by Central Imaging Review Until 18 Weeks After the Start of Treatment
Description: ORR was defined as the percentage of patients who achieved at least one visit response of complete response (CR) or partial response (PR) after the start of treatment. The response criteria evaluation was carried out according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. CR and PR did not need to be confirmed by a subsequent tumor assessment due to blinded central assessment. CR: Disappearance of all target lesions since baseline; PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Tumor assessments were performed prior to trial drug administration, until 18 weeks.
Time Frame: Tumor assessment scans were performed at baseline, Cycle 3 (Week 6), Cycle 5 (Week 12) and at Week 18 ±14 days. Best ORR evaluated until confirmed disease progression, unacceptable toxicity, death or up to 18 weeks, whichever happened earlier.
Population: The FAS contained all randomized patients who received at least 1 dose of trial drug and who had a baseline tumor assessment. Best ORR (CR+PR) is reported for observed values.
Measure: Number; unit: Percentage of patients (%)
Arm/Group | BI 695502 | Avastin® US
Number analyzed (Participants) | 335 | 328
Percentage of patients (%) | 54.0 | 63.1
Statistical Analysis 1: Comparison: BI 695502 vs Avastin® US; Analysis was based on a log-binomial regression model with subsequent transformation of the estimated parameter (ratio of best ORR) respective CIs to the ratio scale. The model included the following explanatory variables: treatment, sex (male versus female), smoking status (never smoked versus current/ex-smoker), NSCLC stage (recurrent versus Stage IV) and ethnicity (East Asian origin versus Non-East Asian); Test type: Equivalence — The null hypothesis was to be rejected in favor of equivalence if the 2-sided 90% confidence interval (CI) for the ratio in best ORR between the treatments was entirely contained within the equivalence margins of 0.736 to 1.359; Log-binomial regression; Ratio of best ORR = 0.8550, 90% CI 2-sided [0.7697 to 0.9506]
Statistical Analysis 2: Comparison: BI 695502 vs Avastin® US; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Additional analysis of the primary endpoint was performed for Japan according to a local protocol amendment Japan. For the submission in Japan, to conclude on equivalence, the 2-sided 95% CI for the ratio of best ORR between the treatments had to be entirely contained within the equivalence margins of 0.736 to 1.359; Log-binomial regression; Ratio of best ORR = 0.8550, 95% CI 2-sided [0.7543 to 0.9700]

2. Secondary Outcome: Percentage of Patients With Selected Treatment-Emergent Adverse Events (TEAEs) For Comparability Assessment of BI 695502 and US-licensed Avastin®
Description: The following selected adverse events (AEs) were evaluated for comparability assessment of BI 695502 and US-licensed Avastin®:
  * Infusion reactions (anaphylactic/hypersensitivity/infusion-related reactions),
  * Thromboembolic events (arterial or venous),
  * Febrile neutropenia,
  * Gastrointestinal perforations,
  * Hypertension,
  * Proteinuria,
  * Pulmonary hemorrhage,
  * Other hemorrhages (not including pulmonary hemorrhages),
  * Wound-healing complications/abscess/fistulas. The analysis of AEs was based on the concept of TEAEs. For non-switched patients, all AEs that started or worsened in severity on or after the first dose of trial drug and prior to the date of last administration of trial medication + 16 weeks inclusive were defined as TEAEs.
Time Frame: From first dose of trial drug until 16 weeks after the last dose of trial medication, up to 218 days.
Population: The Treated Set contained all patients who signed informed consent and who received at least one dose of trial drug.
Measure: Number (95% Confidence Interval); unit: Percentage of patients (%)
Arm/Group | BI 695502 | Avastin® US
Number analyzed (Participants) | 335 | 328
Percentage of patients (%)
  AtLeast 1 AE selected for Comparability Assessment | 52.50 [47.04 to 57.99] | 45.10 [39.65 to 50.68]
  Infusion reactions | 16.70 [12.88 to 21.15] | 13.10 [9.65 to 17.25]
  Thromboembolic events | 6.60 [4.16 to 9.77] | 5.50 [3.28 to 8.53]
  Febrile neutropenia | 3.90 [2.08 to 6.54] | 3.40 [1.69 to 5.92]
  Gastrointestinal perforations | 2.10 [0.84 to 4.26] | 0.60 [0.07 to 2.19]
  Hypertension | 15.50 [11.82 to 19.85] | 16.20 [12.34 to 20.60]
  Proteinuria | 15.80 [12.08 to 20.18] | 14.60 [10.99 to 18.93]
  Pulmonary haemorrhage | 1.20 [0.33 to 3.03] | 0.90 [0.19 to 2.65]
  Other hemorrhages | 20.00 [15.85 to 24.69] | 16.20 [12.34 to 20.60]
  Wound-healing complications/abscess/fistulas | 2.70 [1.24 to 5.04] | 2.10 [0.86 to 4.35]
Statistical Analysis 1: Comparison: BI 695502 vs Avastin® US; At least 1 AE selected for comparability assessment, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.99 to 1.37]
Statistical Analysis 2: Comparison: BI 695502 vs Avastin® US; Infusion reactions, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio (RR) = 1.28, 95% CI 2-sided [0.88 to 1.88]
Statistical Analysis 3: Comparison: BI 695502 vs Avastin® US; Thromboembolic events, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio = 1.20, 95% CI 2-sided [0.64 to 2.32]
Statistical Analysis 4: Comparison: BI 695502 vs Avastin® US; Febrile neutropenia, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.51 to 2.76]
Statistical Analysis 5: Comparison: BI 695502 vs Avastin® US; Gastrointestinal perforations, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio (RR) = 3.43, 95% CI 2-sided [0.79 to 32.82]
Statistical Analysis 6: Comparison: BI 695502 vs Avastin® US; Hypertension, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.66 to 1.39]
Statistical Analysis 7: Comparison: BI 695502 vs Avastin® US; Proteinuria, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.74 to 1.57]
Statistical Analysis 8: Comparison: BI 695502 vs Avastin® US; Pulmonary haemorrhage, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.28 to 10.79]
Statistical Analysis 9: Comparison: BI 695502 vs Avastin® US; Other hemorrhages, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score exact method; Risk Ratio (RR) = 1.24, 95% CI 2-sided [0.88 to 1.74]
Statistical Analysis 10: Comparison: BI 695502 vs Avastin® US; Wound healing complications/ abscesses/ fistulas, risk ratio X (BI 695502) versus Y (US-licensed Avastin®) was defined as (a/(a+b))/(c/(c+d)), where 'a' was the number of patients with TEAEs selected for comparability within treatment group X, 'a+b' was the total number of patients in treatment group X, 'c' was the number of patients with TEAEs selected for comparability within treatment group Y and 'c+d' was the total number of patients in treatment group Y; Test type: Other; Score excat method; Risk Ratio (RR) = 1.26, 95% CI 2-sided [0.47 to 3.57]

3. Secondary Outcome: Progression-Free Survival (PFS) Time as Determined by Investigator Assessment
Description: PFS was defined as the time from randomization until disease progression as determined by Investigator assessment or death from any cause, whichever occurred first during the pre-switch period. Disease progression was assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 millimeters. Tumor assessments were performed prior to trial drug administration. PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumor scans performed at baseline, Cycle 3 (Week 6), Cycle 5 (Week 12), Cycle 7 (Week 18), then every 3 cycles (~9 weeks) until confirmed disease progression. Analysis performed for pre-switch period only; maximum duration of up to 35 cycles (105 weeks).
Population: The Full Analysis Set (FAS) contained all randomized patients who received at least 1 dose of trial drug and who had a baseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BI 695502 | Avastin® US
Number analyzed (Participants) | 335 | 328
Months | 8.34 [7.49 to 8.77] | 9.00 [8.34 to 10.38]
Statistical Analysis 1: Comparison: BI 695502 vs Avastin® US; Analysis based on a Cox-proportional hazards regression model. The model included the following explanatory variables: treatment, sex (male versus female), smoking status (never smoked versus current/ex-smoker), NSCLC stage (recurrent versus Stage IV) and ethnicity (East Asian origin versus non East Asian); Test type: Other; Cox-proportional hazards regression; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [1.02 to 1.45]

4. Secondary Outcome: Overall Survival (OS) Time
Description: OS was defined as the time randomization until death from any cause during the pre-switch period. OS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline until death due to any cause, ie., up to 35 cycles (105 weeks).
Population: The FAS contained all randomized patients who received at least 1 dose of trial drug and who had a baseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BI 695502 | Avastin® US
Number analyzed (Participants) | 335 | 328
Months | 15.57 [14.16 to 17.25] | 19.48 [15.87 to 20.73]
Statistical Analysis 1: Comparison: BI 695502 vs Avastin® US; [analysis description as in outcome 3, analysis 1]; Test type: Other; Cox-proportional hazards regression; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [1.00 to 1.51]

5. Secondary Outcome: Duration of Response (DOR) as Determined by Investigator Assessment
Description: DOR was the time from first documented CR or PR until time of progression as determined by Investigator assessment during the pre-switch period. Tumor assessments were performed prior to trial drug administration. DOR was calculated using the Kaplan-Meier technique.
Time Frame: Tumor scans performed at baseline, Cycle 3 (Week 6), Cycle 5 (Week 12), Cycle 7 (Week 18), then every 3 cycles (~9 weeks) until confirmed disease progression., ie up to 35 cycles (105 weeks).
Population: The FAS contained all randomized patients who received at least 1 dose of trial drug and who had a baseline tumor assessment. Only patients with an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BI 695502 | Avastin® US
Number analyzed (Participants) | 175 | 187
Months | 7.66 [7.03 to 9.03] | 8.94 [7.26 to 10.28]
Statistical Analysis 1: Comparison: BI 695502 vs Avastin® US; [analysis description as in outcome 3, analysis 1]; Test type: Other; Cox-proportional hazards regression; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.88 to 1.48]

ADVERSE EVENTS:
Time Frame: For Pre-switch period: From first dose of trial drug until 112 days (16 weeks) after the last dose of trial medication, up to 218 days. For post-switch period: From the first dose of Avastin® until end of treatment (EOT) visit, up to 127 days.
Groups:
- BI 695502 (Pre-switch): Patients received BI 695502 solution for i.v. infusion, 15 mg/kg bw, every 3 weeks for up to 6 cycles. During the induction cycles, patients also received standard combination chemotherapy consisting of paclitaxel 200 mg/m^2 BSA, followed by carboplatin target AUC 6 mg/mL*min, with adequate pre- and concomitant medication. After Cycle 4 to 6, for responding or stabilized patients, maintenance treatment with BI 695502 monotherapy could be started per the original randomization. Patients then received BI 695502 as a single agent until disease progression, death, withdrawal of consent, unacceptable toxicity, or until the Switch Visit (when each patient was switched to receive commercially available Avastin®), whichever occurred earlier.
- US-licensed Avastin® (Pre-switch): Patients received US-licensed Avastin® solution for i.v. infusion, 15 mg/kg bw, every 3 weeks for up to 6 cycles.
  During the induction cycles, patients also received standard combination chemotherapy consisting of paclitaxel 200 mg/m^2 BSA, followed by carboplatin target AUC 6 mg/mL*min, with adequate pre- and concomitant medication. After Cycle 4 to 6, for responding or stabilized patients, maintenance treatment with US-licensed Avastin® monotherapy could be started per the original randomization. Patients then received US-licensed Avastin® as a single agent until disease progression, death, withdrawal of consent, unacceptable toxicity, or until the Switch Visit (when each patient was switched to receive commercially available Avastin®), whichever occurred earlier.
- BI 695502 (Post-switch): Patients switched from BI 695502 to receive commercially available Avastin®.
- US-licensed Avastin® (Post-switch): Patients switched from US-licensed Avastin® to receive commercially available Avastin®.
Arm/Group | BI 695502 (Pre-switch) | US-licensed Avastin® (Pre-switch) | BI 695502 (Post-switch) | US-licensed Avastin® (Post-switch)
All-Cause Mortality (participants affected / at risk) | 193/335 | 184/328 | 3/42 | 2/46
Serious Adverse Events (participants affected / at risk) | 108/335 | 89/328 | 5/42 | 2/46
Other Adverse Events (participants affected / at risk) | 293/335 | 288/328 | 20/42 | 22/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695502 (Pre-switch) (N=335) | US-licensed Avastin® (Pre-switch) (N=328) | BI 695502 (Post-switch) (N=42) | US-licensed Avastin® (Post-switch) (N=46)
Pneumonia (Infections and infestations) | 9 | 9 | 1 | 0
Lung infection (Infections and infestations) | 2 | 2 | 0 | 0
Peritonitis (Infections and infestations) | 2 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection bacteria (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 11 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 11 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 9 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 5 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Disseminated intravascular coagulati (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 3 | 3 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 6 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 3 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0 | 0
Internal haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Microembolism (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 1 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 1 | 0 | 0
Vascular stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Vasoconstriction (Vascular disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary diseas (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Exposed bone in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 5 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 0
General physical health deterioratio (General disorders) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 5 | 1 | 0 | 0
Platelet count decreased (Investigations) | 2 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial rupture (Cardiac disorders) | 0 | 0 | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagobronchial fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695502 (Pre-switch) (N=335) | US-licensed Avastin® (Pre-switch) (N=328) | BI 695502 (Post-switch) (N=42) | US-licensed Avastin® (Post-switch) (N=46)
Anaemia (Blood and lymphatic system disorders) | 112 | 84 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 61 | 52 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 44 | 47 | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 18 | 23 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 54 | 54 | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 21 | 28 | 0 | 4
Insomnia (Psychiatric disorders) | 15 | 18 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 62 | 59 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 56 | 53 | 0 | 1
Headache (Nervous system disorders) | 26 | 25 | 1 | 2
Paraesthesia (Nervous system disorders) | 20 | 19 | 0 | 0
Dysgeusia (Nervous system disorders) | 13 | 17 | 0 | 0
Hypertension (Vascular disorders) | 49 | 51 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 32 | 0 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 | 32 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 31 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 | 10 | 0 | 1
Nausea (Gastrointestinal disorders) | 73 | 75 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 60 | 45 | 1 | 1
Vomiting (Gastrointestinal disorders) | 56 | 37 | 1 | 1
Constipation (Gastrointestinal disorders) | 51 | 44 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 155 | 149 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 17 | 16 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 35 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 38 | 29 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 14 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 | 10 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 18 | 1 | 0
Proteinuria (Renal and urinary disorders) | 51 | 46 | 8 | 6
Fatigue (General disorders) | 54 | 53 | 2 | 1
Asthenia (General disorders) | 22 | 29 | 1 | 2
Malaise (General disorders) | 19 | 13 | 0 | 0
Pyrexia (General disorders) | 17 | 21 | 0 | 1
Platelet count decreased (Investigations) | 41 | 33 | 0 | 0
Neutrophil count decreased (Investigations) | 39 | 42 | 0 | 0
White blood cell count decreased (Investigations) | 30 | 19 | 0 | 0
Alanine aminotransferase increased (Investigations) | 24 | 32 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 22 | 31 | 1 | 6
Weight decreased (Investigations) | 21 | 22 | 2 | 1
Blood cholesterol increased (Investigations) | 20 | 16 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 19 | 30 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 17 | 25 | 0 | 3
Haemoglobin decreased (Investigations) | 5 | 17 | 0 | 0

LIMITATIONS AND CAVEATS:
From 21 December 2017, after Week 18 primary analysis data cut-off, the Sponsor recommended to switch patients from BI 695502/US-licensed Avastin® to Avastin®. The main analyses to report all endpoint and AE results was the pre-switch period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT02272413/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT02272413/SAP_001.pdf